CLINICAL TRIAL: NCT02489032
Title: Web-Based Training for EAP Alcohol Screening, Brief Intervention, and Refer
Acronym: BigAl2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BIG Al 2; 2R44AA021053 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Alcohol Consumption; Alcohol Abuse
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBIRT Training & Support Tool (Experimental): The SBIRT Training & Support Tool has two components, both of which will be evaluated: (1) online SBIRT Training for EAP and behavioral health practitioners conducting alcohol SBIRT with their adult clients and (2) mobile/web interactive alcohol screening tools and brief intervention protocols to facilitate use of SBIRT by practitioners.
  Interventions: Behavioral: SBIRT Training & Support Tool
- Waitlist control (Other): Subjects randomized to the control condition will be placed on a wait-list and given access to the SBIRT Training & Support Tool after 3 months and completion of the 3-month follow-up assessment.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: SBIRT Training & Support Tool — Program to train EAP/behavioral health practitioners in conducting alcohol SBIRT
  Arms: SBIRT Training & Support Tool
Other: Waitlist Control — 3-month wait-list and then provided access to the SBIRT training program
  Arms: Waitlist control

SUMMARY:
The goal of the proposed research is to complete the development of a web-based program to train Employee Assistance Program (EAP) and EAP-affiliated managed behavioral health organization (MBHO) practitioners to conduct screening, brief intervention, and referral to treatment (SBIRT) for problem alcohol use among working adults.

DETAILED DESCRIPTION:
In Phase 2, the investigators propose to develop the SBIRT Training & Support Tool with two components: (1) online SBIRT Training for call-center and face-to-face practitioners conducting alcohol SBIRT and (2) SBIRT Support Tool with mobile/web interactive alcohol screening tools and brief intervention protocols to facilitate use of SBIRT by practitioners. The SBIRT Training component will provide practitioners with the skills, knowledge, motivation, and self-efficacy to: (a) screen their clients for unhealthy alcohol use with validated screening tools; (b) provide brief, motivational interviewing-informed intervention; and (c) make appropriate referrals. The training program will incorporate the Phase 1 content and expand the curriculum to include the use of additional validated alcohol screening tools. Content for alcohol SBIRT will be derived from NIAAA evidence-based materials.

The SBIRT Support Tool will provide a mobile/web interface for practitioners to use interactive screening and brief intervention forms with (a) prompts for validated questions in the screening or brief intervention; (b) motivational interviewing-informed dialogue suggestions; (c) online resources (i.e., standard drink list; importance, confidence rulers); and (d) alcohol education and referral information. The practitioner will use the SBIRT Support Tool to (a) screen clients for alcohol use with interactive validated screening tools; (b) provide brief intervention for individuals based on their screening score; and (c) provide referral to treatment for individuals based on their screening score.

ELIGIBILITY:
Inclusion Criteria:

* EAP/BH practitioners will be employed at an EAP or behavioral health organization
* have an e-mail account
* access to high-speed Internet connection
* speak and read English

Exclusion Criteria:

* younger than 18
* not an EAP practitioner
* no access to e-mail
* no access to the Internet
* do not speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2016-11-13 (Actual)

PRIMARY OUTCOMES:
SBIRT implementation | 3 months
  Situation judgment tests (SJT) will assess trainee's responses to real-life situations and behaviors. The SJT will consist of 9 brief (20-30 seconds) audio-based vignettes of motivational interviewing and alcohol SBIRT in typical clinical and counseling situations. For each of the 9 SJTs, trainees will identify MI/SBIRT-compliant responses.

SECONDARY OUTCOMES:
Perceived Competence | 3 months
  13-item scale assessing trainee's perceived competence (self-efficacy) for using motivational interviewing and alcohol SBIRT skills
Knowledge | 3 months
  23-item scale assessing trainee's knowledge of motivational interviewing and alcohol SBIRT concepts
Attitudes | 3 months
  10-item scale assessing trainee's attitudes about conducting motivational interviewing and alcohol SBIRT with clients

CONTACTS AND LOCATIONS:
Overall Officials: Amelia J Birney, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science

IPD SHARING:
Plan to Share IPD: No